CLINICAL TRIAL: NCT01488656
Title: Effect of an Antioxidant and Anti-inflammatory Dietary Supplement Pack on the Adverse Physiological Actions Associated With Acute PM2.5 Exposure
Brief Title: Effects of Dietary Supplements on Response to Air Pollution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Utah State University (Other)
Collaborators: USANA Health Sciences (Industry)
Responsible Party: Principal Investigator, Michael Lefevre, USTAR Professor, Utah State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: USU #4001; 4011 (Other Grant/Funding Number: USANA Health Sciences)
Record Dates: First submitted 2011-12-06; First posted 2011-12-08 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Inflammation
Keywords: Antioxidants; Dietary supplements; Forced vital lung capacity; Exhaled nitric oxide; Air pollution
MeSH Terms: conditions — Inflammation | interventions — Antioxidants

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo dietary supplements (Placebo Comparator): Visually identical inactive dietary supplement pack
  Interventions: Dietary Supplement: Placebo
- Active dietary supplements (Experimental): Combination of antioxidants, minerals, fish oil, proflavanol and vitamin D
  Interventions: Dietary Supplement: Antioxidant, anti-inflammatory dietary supplement

INTERVENTIONS:
Dietary Supplement: Placebo — 7-pill placebo dietary packed visually identical to active dietary supplement
  Arms: Placebo dietary supplements
Dietary Supplement: Antioxidant, anti-inflammatory dietary supplement — A combination of dietary supplements including: β-carotene, vitamin C, vitamin D3, vitamin E, vitamin K, thiamin, riboflavin, niacin, vitamin B6, folate, vitamin B12, biotin, pantothenic acid, calcium, iodine, magnesium, zinc, selenium, copper, manganese, chromium, molybdenum, boron, silicon, vanadium, eicosapentaenoic acid, docosahexaenoic acid, olive extract, mixed tocopherols, bioflavonoids, inositol, choline, N-acetyl L-cysteine, bromelain, coenzyme Q10, turmeric extract, lutein, lycopene, broccoli concentrate, grape seed extract
  Other Names: USANA Mega Antioxidant; USANA Chelated Mineral; USANA Proflavanol C 200; USANA Vitamin D
  Arms: Active dietary supplements

SUMMARY:
This study will determine if a comprehensive antioxidant/anti-inflammatory dietary supplement pack can offer protection against a decline in lung function and increase in inflammation and oxidative stress following acute exposure to particulate matter air pollution with a diameter <2.5 µm (PM2.5).

The investigators hypothesis is a follows: Compared to an appropriate control, supplementation with a comprehensive antioxidant/anti-inflammatory dietary supplement pack for 18 weeks will: 1) reduce the decline in lung function following acute exposure to naturally occurring elevations in PM2.5 levels as measured by exhaled nitric oxide levels and forced vital lung capacity; and 2) reduce changes in pro-inflammatory cytokines following acute exposure to naturally occurring elevations in PM2.5 levels as measured by plasma levels of C-reactive protein.

DETAILED DESCRIPTION:
The study will be conducted in Cache County, UT. Surrounded by tall mountains (2513-3042 m), and subject to frequent winter atmospheric inversions characterized by stagnant air that traps and concentrates pollutants, Cache Valley, home to 120,000 inhabitants, is particularly susceptible to high particulate air pollution during the winter months.

A total of 70 individuals (with the goal of completing 60) between the ages of 45-80 will be recruited from Cache County, UT. Eligible participants will be randomly assigned to one of two treatment arms (Placebo Dietary Supplements, Active Dietary Supplements) in a manner to provide balanced assignment between the two arms with respect to age, sex and baseline exhaled nitric oxide levels.

Participants assigned to the Placebo or Active arms will be provided with sealed envelopes or bottles containing dietary supplements (or matched placebos) along with instructions as to when to consume the supplements. Participants will be instructed to consume their supplements twice a day with meals containing a small amount of fat (at least 3 grams) in order to optimize the absorption of fat soluble nutrients. They will also be instructed to consume the supplements with liquids in order to enhance absorption and to minimize GI upset and choking potential. Participants will be asked to maintain their typical diet for the 18 weeks of the study.

Routine Clinic Visits are scheduled at two week intervals for the length of the study (with accommodations made for Holiday schedules). During these visits, participants will: 1) receive a sufficient supply of supplements to last until the next routine clinic visit; 2) return any unused supplements; 3) be provided an opportunity to describe any adverse events/reactions to the supplements; 4) describe any health issues experienced since the previous exam; and 5) have their weight and blood pressure assessed.

Endpoint Clinic Visits are scheduled to coincide with low and high PM2.5 exposure. Starting on Jan 2, participants will be notified of a potential endpoint assessment day when the PM2.5 levels are predicted by the Utah Department of Environmental Quality, Division of Air Quality, to rise above 30 µg/m3 (peak event) or fall below 8 µg/m3 (baseline event). Endpoint visits will take place 24 hrs following these peak and baseline events. Based on historical patterns, we anticipate at least three peak events, with corresponding baseline assessments, during the intervention time period. For purposes of analysis, each peak event will be paired with the nearest baseline event so that both events are captured at a similar time after initiation of the intervention.

At each endpoint clinic visit, participants will undergo assessments of lung function and systemic inflammation. Blood samples will be obtained for potential future analysis of additional markers of systemic inflammation and plasma antioxidant capacity.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of any race or ethnicity
* Body Mass Index (BMI) between 19 - 34 kg/m2
* Non-smoking status
* Willing to consume assigned dietary supplements for 18 weeks.

Exclusion Criteria:

* BMI <19 or >34 kg/m2
* Uncontrolled hypertension defined as diastolic blood pressure >=95 mm Hg or systolic blood pressure >=160 mm Hg
* Documented presence of atherosclerotic disease and/or cardiopulmonary disease
* History of frequent falls
* History of drug or alcohol abuse
* History of unstable depression or mental illness within the last 6 months for which the PI believes could impact the participant's ability to comply with study requirements
* Unwilling to discontinue use of conventional multivitamin/mineral or other supplements at least two weeks prior to the study start
* Participating in or planning to begin a weight loss diet during the study period
* Chronic use of over-the-counter medication which would interfere with study endpoints including NSAIDS, laxatives and antacids
* Difficulty in swallowing pills
* Lifestyle or schedule incompatible with the study protocol

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2011-11; Primary Completion 2012-03 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Forced vital lung capacity (FVC) | Six times over 3 months to coincide with high and low PM2.5 exposure

SECONDARY OUTCOMES:
Forced expiratory volume in first second (FEV1) | Six times over 3 months to coincide with high and low PM2.5 exposure
Fractional exhaled nitric oxide (FeNO) | Six times over 3 months to coincide with high and low PM2.5 exposure
C-reactive protein | Six times over 3 months to coincide with high and low PM2.5 exposure

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lefevre, PhD, Principal Investigator — Utah State University